CLINICAL TRIAL: NCT00714688
Title: A Multicentre, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Response Study to Evaluate Efficacy and Safety of Prolonged Release (PR) OROS Methylphenidate (54 and 72 mg/Day) in Adults With Attention Deficit/Hyperactivity Disorder
Brief Title: A Study to Evaluate Effectiveness and Safety of Prolonged Release OROS Methylphenidate in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014566; 42603ATT3013
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2010-04-21 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Attention Deficit/ Hyperactivity Disorder
Keywords: Adult; ADHD; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): prolonged release (PR) OROS methylphenidate 54 mg 18+36mg once daily for 13 weeks
  Interventions: Drug: prolonged release (PR) OROS methylphenidate 54 mg
- 002 (Experimental): prolonged release (PR) OROS methylphenidate 72 mg 2x36mg once daily for 13 weeks
  Interventions: Drug: prolonged release (PR) OROS methylphenidate 72 mg
- 003 (Placebo Comparator): Placebo 2xplacebo once daily for 13 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: prolonged release (PR) OROS methylphenidate 54 mg — 18+36mg once daily for 13 weeks
  Arms: 001
Drug: prolonged release (PR) OROS methylphenidate 72 mg — 2x36mg once daily for 13 weeks
  Arms: 002
Drug: Placebo — 2xplacebo once daily for 13 weeks
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the efficacy of 2 fixed dosages of Prolonged Release (PR) OROS methylphenidate (54 and 72 mg/day) compared with placebo in adult patients with attention deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of 2 fixed dosages of Prolonged Release (PR) OROS methylphenidate (54 and 72 mg/day) compared with placebo in adult patients with attention deficit/hyperactivity disorder (ADHD). The primary efficacy criterion will be the change in the sum of the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated Conners' Adult ADHD Rating Scale (CAARS), from start of treatment to the end of the double-blind treatment. Hypothesis of the primary objective states that either PR OROS methylphenidate dose is more effective than placebo after 13 weeks of treatment in adult patients with ADHD. This is a multicentre, double-blind, randomized, placebo-controlled, parallel group, dose-response study. Patients will be randomized into one of 3 treatment groups to receive oral dosages of PR OROS methylphenidate 54 or 72 mg, or placebo once daily. The study includes a treatment period of 13 weeks. Patients will be titrated from a starting dose of 36 mg/day for 7 days, to 54 or 72 mg/day at Day 8, after which treatment will be administered for 12 weeks. The study will include a screening period of up to 2 weeks, during which current therapy, not allowed during the study can be tapered down and discontinued (with the exception of fluoxetine or MAO (monoamine oxidase) inhibitors for which a maximum screening period of 4 weeks will be allowed). A post-study visit for collection of additional efficacy and safety data will be scheduled for one week after a patient's final dose of study drug. Adults with a diagnosis of ADHD according to DSM-IV criteria with some symptoms before age 7 years that continue to meet these criteria at the time of assessment will be enrolled in this study. ADHD is not diagnosed if the symptoms are better accounted for by another psychiatric disorder (e.g. mood disorder, anxiety disorder, psychotic disorder, personality disorder). The patient (and if possible, informant) must also describe a chronic course of ADHD symptomatology from childhood to adulthood. The description of this chronic course can be patient-based and previous documented diagnosis and/or treatment is not required. Approximately 300 patients (100 in each randomized treatment group) will participate in this study. The primary efficacy criterion will be the change in the sum of the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated CAARS from baseline to the end of treatment (end of 13 weeks or last post-baseline assessment). This variable will be compared between each dosage group and placebo using an ANCOVA model. Other end points will include changes from baseline to the end of the treatment in the CAARS subscales and assessment of the clinical global impression - global change subscale (CGI-C). Onset of therapeutic effect and responder rate will also be determined. In addition, morning / evening (8 pm) CAARS-S:S assessments will be performed at baseline and on Days 34, 35, 90 and 91. Safety evaluations will include monitoring of adverse events (AEs), clinical laboratory tests (hematology; biochemistry), pregnancy testing, vital signs (supine and standing blood pressure, pulse) and weight, ECG. Patients will be randomized to receive PR OROS methylphenidate 54 or 72 mg, or placebo once daily. Study drug will be administered daily in the morning for up to 13 weeks. Since there is no food effect with methylphenidate, drug administration can be under fed or fasted conditions. Patients will start at a dosage of 36 mg. At Week 2, patients will receive 54 or 72 mg PR OROS methylphenidate for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV) and confirmed by the Conners' Adult ADHD Diagnostic Interview for DSM IV
* Described chronic course of ADHD symptomatology from childhood to adulthood, with some symptoms present before age 7 years and continue to meet DSM-IV criteria at the time of assessment
* CAARS score of at least or equal to 24 as determined by investigator at screening visit
* Patient agrees to take only the supplied study drug as treatment for ADHD during the study
* Patient agrees not to initiate a new behavioral modification program during the study or if currently using a behavioral modification program agrees not to change this program during the study.

Exclusion Criteria:

* Known to be a non-responder to methylphenidate, or patient has a child known to be a non-responder to methylphenidate
* Has been treated with any methylphenidate-containing medication within 1 month of screening visit
* Participation in and premature withdrawal from 42603ATT3002, CR002479 or 42603ATT3004, CR011068 study
* Known allergy or hypersensitivity to methylphenidate, or components of PR OROS methylphenidate
* Any clinically unstable psychiatric condition including, but not limited to the following: acute mood disorder, bipolar disorder, acute obsessive-compulsive disorder (OCD), anti-social personality disorder, borderline personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (42):
- Belgium (5):
  - Antwerp
  - Brussels
  - Kortenberg
  - Mechelen
  - Mons
- Denmark (3):
  - Aarhus
  - Hjørring
  - Holstebro
- Finland (3):
  - Helsinki
  - Oulu
  - Pori
- France (3):
  - Montpellier
  - Nice
  - Paris
- Germany (10):
  - Ahrensburg
  - Aschaffenburg
  - Berlin
  - Düsseldorf
  - Essen
  - Freiburg im Breisgau
  - Mannheim
  - München
  - Saarbrücken
  - Würzburg
- Netherlands (2):
  - Nijmegen
  - The Hague
- Norway (4):
  - Bryne
  - Oslo
  - Ottestad
  - Skien
- Spain (2):
  - Barcelona
  - Madrid
- Sweden (6):
  - Huddinge
  - Linköping
  - Lund
  - Malmo
  - Örebro
  - Uppsala
- Switzerland (2):
  - Basel Bs
  - Zurich
- United Kingdom (2):
  - Cambridge
  - Swansea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 4 February 2008 (first subject in) to 2 April 2009 (last subject out).
Pre-assignment Details: After enrolment patients entered a screening period of up to 2 weeks included the tapering and discontinuation of current forbidden treatment (except if fluoxetine or Monoamine Oxidase (MAO) inhibitors needed to be tapered, in which case a screening period of 4 weeks was allowed).
Groups:
- Placebo: 2 tablets placebo once daily for 13 weeks
- 54 mg PR OROS MPH: Prolonged-release (PR) OROS methylphenidate 18 + 36 mg once daily for 13 weeks
- 72 mg PR OROS MPH: Prolonged-release (PR) OROS methylphenidate 2 tablets 36 mg once daily for 13 weeks
Period: Overall Study
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Started | 97 | 90 | 92
Completed | 68 | 55 | 55
Not Completed | 29 | 35 | 37
Not completed — Lack of Efficacy | 14 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Lost to Follow-up | 5 | 2 | 0
Not completed — Adverse Event | 2 | 15 | 19
Not completed — Subject Non-compliant | 3 | 5 | 5
Not completed — Ineligible to Continue the Study | 0 | 1 | 1
Not completed — Sponsor's Decision | 0 | 2 | 0
Not completed — Other | 1 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH | Total
Number analyzed (Participants) | 97 | 90 | 92 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 4
  Between 18 and 65 years | 96 | 89 | 90 | 275
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.81) | 35.8 (11.71) | 35.8 (10.08) | 35.7 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 42 | 133
  Male | 52 | 44 | 50 | 146

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit/Hyperactivity Disorder (ADHD) Symptoms Total Score of the Conners Adult ADHD Rating Scale (CAARS)
Description: The primary endpoint was the change in the ADHD symptoms total score of the investigator-rated CAARS from baseline to the last assessment in the double-blind treatment period. CAARS assesses ADHD symptoms and behaviors in adults using a scale ranging from 0 (best) to 54 (worst). For subjects without a post-baseline efficacy measurement, a change of 0 units was imputed.
Time Frame: from baseline to 13 weeks
Population: The ITT analysis set (includes all randomized subjects) was considered the primary efficacy analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Number analyzed (Participants) | 97 | 90 | 92
units on a scale
  Baseline | 36.5 (6.05) | 35.6 (6.75) | 37.3 (6.35)
  Endpoint | 26.1 (10.59) | 23.0 (11.07) | 21.6 (10.21)
  Change at Endpoint | -10.4 (11.03) | -12.5 (10.38) | -15.7 (10.80)
Statistical Analysis 1: Comparison: Placebo vs 54 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p = 0.136, ANCOVA — The p value was adjusted for multiplicity via Dunnett's test procedure; Treatment, gender and country were used as factors and baseline value and age were used as covariates; Difference in Least-Squares Means = -2.7, 95% CI [-6.04 to 0.67], Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: Placebo vs 72 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p = 0.002, ANCOVA — The p value was adjusted for multiplicity via Dunnett's test procedure; Treatment, gender and country were used as factors and baseline value and age were used as covariates; Difference in Least-Squares Means = -4.9, 95% CI [-8.22 to -1.55], Standard Error of Mean 1.50

2. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) From Baseline to End of Treatment
Description: The CGI-S rating scale is used to rate the severity of a subject's illness on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe illness). The change in CGI-S was assessed from baseline to end of treatment (week 13 or or last post-baseline assessment)
Time Frame: from baseline to13 weeks
Population: The ITT analysis set (includes all randomized subjects) was considered the primary efficacy analysis set.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Number analyzed (Participants) | 97 | 90 | 92
units on a scale | 0.0 [-6 to 1] | -1.0 [-4 to 1] | -1.0 [-4 to 1]
Statistical Analysis 1: Comparison: Placebo vs 54 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p = 0.216, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; The ANCOVA model was performed on ranked data. Treatment, gender & country were used as factors and baseline value & age were used as covariates
Statistical Analysis 2: Comparison: Placebo vs 72 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; The ANCOVA model has been performed on ranked data. Treatment, gender & country were used as factors and baseline value & age were used as covariates

3. Secondary Outcome: Clinical Global Impression-Change (CGI-C)
Description: The CGI-C rating scale is used to rate the change in severity of the subject's illness compared to baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: 13 weeks
Population: The ITT analysis set (includes all randomized subjects) was considered the primary efficacy analysis set.It excludes patients for which either a baseline or end of treatment value was missing.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Number analyzed (Participants) | 93 | 84 | 92
units on a scale | 3.0 [1 to 6] | 2.5 [1 to 5] | 2.0 [1 to 6]
Statistical Analysis 1: Comparison: Placebo vs 54 mg PR OROS MPH; Test type: Superiority or Other; p = 0.052, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; The ANCOVA model has been performed on ranked data. Treatment, gender and country were used as factors and age was used as a covariate
Statistical Analysis 2: Comparison: Placebo vs 72 mg PR OROS MPH; Test type: Superiority or Other; p = 0.002, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Change in Conners Adult ADHD Rating Scale Self Report Short Version (CAARS-S:S) Total Score
Description: The CAARS-S:S is a 26-item self-report scale that measures symptoms based on the DSM-IV criteria for ADHD. Respondents were asked to rate items pertaining to their behavior/problems using the following 4-point scale (from 0 = Not at all, never; to 3 = Very much, very frequently). The CAARS-S:S total score range is from 0 (best) to 78 (worse). The change in CAARS-S:S was assessed from baseline to end of treatment (week 13 or or last post-baseline assessment)
Time Frame: from baseline to 13 weeks
Population: The ITT analysis set (includes all randomized subjects) was considered the primary efficacy analysis set. It excludes patients for which a baseline value was missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Number analyzed (Participants) | 94 | 85 | 90
units on a scale | -8.5 (11.64) | -12.8 (13.42) | -12.6 (13.84)
Statistical Analysis 1: Comparison: Placebo vs 54 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p = 0.023, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; Treatment, gender and country were used as factors and baseline value and age were used as covariates; Difference in Least-Squares Means = -4.2, Standard Error of Mean 1.86
Statistical Analysis 2: Comparison: Placebo vs 72 mg PR OROS MPH; Statistical analysis of change from baseline at endpoint; Test type: Superiority or Other; p = 0.016, ANCOVA — Comparison with placebo was performed without multiplicity adjustment; Treatment, gender and country were used as factors and baseline value and age were used as covariates; Difference in Least-Squares Means = -4.4, Standard Error of Mean 1.83

ADVERSE EVENTS:
Description: All safety parameters were analyzed using the safety analysis set (ie all subjects who were randomized and received at least 1 dose of study medication). One subject (54mg) in the ITT analysis set was randomized but not treated. Therefore, this subject was not included in the safety analysis set.
Arm/Group | Placebo | 54 mg PR OROS MPH | 72 mg PR OROS MPH
Serious Adverse Events (participants affected / at risk) | 2/97 | 3/89 | 2/92
Other Adverse Events (participants affected / at risk) | 56/97 | 72/89 | 79/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | 54 mg PR OROS MPH (N=89) | 72 mg PR OROS MPH (N=92)
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis Infective (Infections and infestations) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | 54 mg PR OROS MPH (N=89) | 72 mg PR OROS MPH (N=92)
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 17 | 26
Anorexia (Metabolism and nutrition disorders) | 4 | 6 | 12
Insomnia (Psychiatric disorders) | 11 | 13 | 15
Initial Insomnia (Psychiatric disorders) | 2 | 7 | 9
Agitation (Psychiatric disorders) | 1 | 2 | 8
Anxiety (Psychiatric disorders) | 4 | 8 | 8
Depressed Mood (Psychiatric disorders) | 5 | 4 | 6
Restlessness (Psychiatric disorders) | 0 | 8 | 3
Headache (Nervous system disorders) | 25 | 25 | 27
Dizziness (Nervous system disorders) | 6 | 5 | 11
Tremor (Nervous system disorders) | 1 | 5 | 4
Dry Mouth (Gastrointestinal disorders) | 3 | 12 | 20
Nausea (Gastrointestinal disorders) | 8 | 15 | 16
Weight Decreased (Investigations) | 4 | 9 | 17
Heart Rate Increased (Investigations) | 0 | 4 | 6
Tachycardia (Cardiac disorders) | 0 | 6 | 10
Palpitations (Cardiac disorders) | 0 | 7 | 7
Fatigue (General disorders) | 4 | 3 | 9
Irritability (General disorders) | 6 | 5 | 2
Nasopharyngitis (Infections and infestations) | 14 | 13 | 11
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4

LIMITATIONS AND CAVEATS:
Study was not designed to statistically compare the 54 mg with the 72 mg dose. Study medication was not titrated to the assigned dose as in clinical practice. This could have differentially affected treatment emergence of AEs and patient retention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days